CLINICAL TRIAL: NCT04013828
Title: Recurrent High-grade Glioma: Experiences of Patients and Their Close Relatives During the Treatment Decision-making Process.
Brief Title: Treatment Decision-making in Patients With Recurrent High-grade Glioma
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Region of Southern Denmark (Other); Danish Cancer Society (Other); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Helle Sørensen von Essen, Principal Investigator, Odense University Hospital
Other Study IDs: OP870
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Malignant Glioma; Life Experiences
Keywords: High-grade glioma; Patient experiences; Decision-making; Patient involvement
MeSH Terms: conditions — Glioma; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with recurrent high-grade glioma
- Relatives: Close relatives of patients with recurrent high-grade glioma

SUMMARY:
This qualitative study explores the lived experience of high-grade glioma patients and their close relatives at time of recurrence. With focus on the decision-making about treatment and care..

DETAILED DESCRIPTION:
High-Grade Glioma is a life-threatening disease that can cause the patient substantial physical, mentally and psychosocially impairment. The life expectancy is short, and a majority of patients experience recurrence of tumour growth. At time of recurrence, the treatment possibilities can include surgery, oncological treatment and/or palliative care.

In this situation the patients and their close relatives need to make a difficult balancing between benefits and trade offs.

Little is known about how the patients and their close relatives experience the recurrence and the decision-making process.

The objective of this study is therefore to explore the perspectives, experiences and needs in patients and their close relatives in relation to the decision-making process at time of recurrence.

Data will be generated through semi-structured interviews. Interviews will be analysed and interpreted using a Ricoeur inspired method of qualitative analysis.

The study is part of a larger PhD-study.

ELIGIBILITY:
Inclusion Criteria:

* The patient is offered surgical treatment (after an assesment done by the multidisciplinary team)
* Able to speak and understand danish
* Able to participate in an interview
* Able to give informed concent for participation

Exclusion Criteria:

* Patients with severe cognitive impairment which prohibits them from either giving informed concent or participating in interview.
* Relatives are excluded if the patient do not give concent for the participation of relatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two study populations:
  1. - Adult patients with recurrence of high-grade glioma who are offered surgical treatment as one of the treatment possibilities.
  2. - The adult relative most involved in the decision-making. The relative is apointed by the patient and the patient gives written concent to the relative' participation.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Experiences of patients and relatives | Interviews are performed 2-6 weeks after the decision-making
  How patients and their close relatives experience the decision-making process
Involvement preferences | Interviews are performed 2-6 weeks after the decision-making
  The preferences of patients and relatives for being involved in the decision-making.

CONTACTS AND LOCATIONS:
Overall Officials: Frantz Rom Poulsen, Professor, Study Director — Department of Neurosurgery Odense University Hospital DK-5000 Odense C DENMARK
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital; Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No